CLINICAL TRIAL: NCT04204226
Title: Assessing the Feasibility, Acceptability, and Preliminary Efficacy of an Adaptive Intervention Approach for Children With Autism and Disruptive Behavior: A Pilot Study
Brief Title: Autism and Disruptive Behavior Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eagles Autism Challenge, Inc (Unknown); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-016364
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: ASD; Child Behavior Problem
Keywords: Autism spectrum disorder; Sequential Multiple Assignment Randomized Trial
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Social Work

STUDY DESIGN:
Intervention Model Description: Study Phase 1- Children with autism spectrum disorder (ASD) and disruptive behavior will be randomized to social work (SW) or autism behavioral health navigation (ABHN) Study Phase 2- Children who are responding to their Phase 1 intervention will remain in that intervention; children who are not responding to their Phase 1 intervention in the social work arm will be randomly assigned to either ABHN or ABHN+Complex Autism Program (CAP). Those not responding in the ABHN arm will receive ABHN + CAP.
Who Masked: Participant
Masking Description: Given the nature of the intervention families will not be blind to the intervention they are receiving. During phase 1 the investigator providing the clinical global impression (CGI) scores will be blind to the child's group assignment. Families will be asked not to discuss their work with a social worker or ABHN when completing interview questions at the interim assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Worker vs Autism Behavioral Health Navigation (ABHN) (Experimental): Phase 1: Families providing informed consent will then be randomized to social work consultation or to the Autism Behavioral Health Navigation (ABHN) intervention.
  Non-responders to ABHN will move to ABHN + Complex Autism Program (CAP).
  Interventions: Behavioral: Social Worker; Behavioral: Autism Behavioral Health Navigation (ABHN)
- Social work + ABHN vs Social work + ABHN + CAP (Experimental): At 3 months, children who are considered to be "responders" to their current treatment will continue; children who are "nonresponders" in the social work arm of the study will be randomized to either ABHN or ABHN+CAP. Children in the ABHN arm who are non-responders will receive ABHN + CAP
  Interventions: Behavioral: Social work + ABHN; Behavioral: Social work + ABHN + CAP

INTERVENTIONS:
Behavioral: Social Worker — The social worker will discuss the clinician's recommendations for needed services and how to access the services. The family will be provided the social worker's contact information and be encouraged to reach out with more questions or if more information is needed.
  Arms: Social Worker vs Autism Behavioral Health Navigation (ABHN)
Behavioral: Autism Behavioral Health Navigation (ABHN) — The goal of the ABHN intervention is to ensure access to recommended community behavioral health services, decrease parent stress levels, and/or improve child sleep and activity levels in order to reduce disruptive behaviors. Navigators will check-in at least weekly by telephone, email, or text message (as per family preference) during the first 4 weeks of the intervention and at least every 2 weeks for the remainder of the intervention or until ABHN and family agree that all goals and action steps in the Family Care Plan are completed.
  Arms: Social Worker vs Autism Behavioral Health Navigation (ABHN)
Behavioral: Social work + ABHN — After 3 months, children whose ABC Irritability Subscale scores improve by less than 5 points who received the social work intervention can be randomized to ABHN
  Arms: Social work + ABHN vs Social work + ABHN + CAP
Behavioral: Social work + ABHN + CAP — After 3 months, children whose ABC Irritability Subscale scores improve by less than 5 points who received the social work intervention can be randomized to ABHN+Complex Autism Program (CAP)
  Arms: Social work + ABHN vs Social work + ABHN + CAP

SUMMARY:
Investigators seek to transform the delivery of health care to children with autism spectrum disorder (ASD) and behavioral health problems (and their families) by developing an innovative tiered set of interventions. Investigators aim to demonstrate that for children with ASD and disruptive behavior a family navigation-based intervention (autism behavioral health navigation; ABHN) will be feasible and more acceptable to families than brief social work consultation. For children with persistent disruptive behavior despite the social work or ABHN intervention Investigators will evaluate the feasibility and acceptability of adding consultation with an interprofessional team of ASD experts.

DETAILED DESCRIPTION:
Context: It is often challenging to help families of children with autism spectrum disorder (ASD) manage disruptive behaviors. Family navigation and interprofessional care are promising care strategies that could be applied to care for these children.

Objectives: Investigators aim to demonstrate that for children with ASD and disruptive behavior a family navigation-based intervention (autism behavioral health navigation; ABHN) will be feasible and more acceptable to families than brief social work consultation. For persistent disruptive behavior despite the social work or ABHN intervention we will evaluate the feasibility and acceptability of adding consultation with an interprofessional team of ASD experts (Complex Autism Program; CAP).

Study Design: Investigators will conduct a Sequential Multiple Assignment Randomized Trial (SMART) of social work consultation, ABHN, and ABHN+CAP.

Setting/Participants:Participants will be children age 5-12 years, diagnosed with an ASD, receiving care for ASD at the Children's Hospital of Philadelphia (CHOP) in the Division of Developmental and Behavioral Pediatrics (DBP), Division of Neurology, or in the Department of Child and Adolescent Psychiatry and Behavioral Sciences (DCAPBS), and exhibiting high levels of disruptive behaviors (defined as an elevated score on the Aberrant Behavior Checklist (ABC) Irritability subscale and an elevated score on the Clinical Global Impression - Severity (CGI-S)). A parent of the child involved in coordinating the child's care will also be a participant in the study.

Study Interventions and Measures: Interventions include brief social work consultation, ABHN, and an interprofessional evaluation. The primary outcome measure will be the Aberrant Behavior Checklist (ABC) Irritability subscale. Secondary measures include the Clinical Global Impression - Severity and Clinical Global Impression - Improvement (CGI-S and CGI-I), parent ratings of child behavior, parenting stress, and measures of feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

1. Child is age 5 through 12 years 11 months
2. Diagnosed with autism spectrum disorder (ASD) and receives care for ASD at the Children's Hospital of Philadelphia (CHOP) in Developmental and Behavioral Pediatrics (DBP) or Child Neurology, or in Department of Child and Adolescent Psychiatry and Behavioral Sciences (DCAPBS)
3. Child exhibits disruptive behaviors characterized by tantrums, outbursts, self-injurious, or aggressive behaviors with a Clinical Global Impression severity (CGI-S) for the disruptive behavior of at least 4
4. A caregiver completed Aberrant Behavior Checklist (ABC-2) Irritability subscale score is greater than 13
5. A parent of the child who is involved in coordinating the child's care will also participate as a research subject.

Exclusion Criteria:

1. Child requires crisis intervention or urgent psychiatric consultation
2. Referring physician or psychologist will not be providing ongoing management of the child's behavioral challenges.
3. Parent needs a different intervention or type of assistance than will be available through the study
4. Families who live outside a 40 mile radius from the Children's Hospital of Philadelphia (CHOP -main)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Number of children referred to the study each month meeting eligibility requirements | 9 months
  Prescribing clinicians from the following Divisions and Departments (DBP, Neurology, DCAPBS) will refer patients age 5-12 with ASD and disruptive behavior to the study. The number of children referred will be determined by counting the participants in the study who meet the inclusion criteria.

SECONDARY OUTCOMES:
Number of families successfully contacted by the navigator or social worker | 9 months
  The number of families successfully contacted will be determined by reviewing contact logs of all contacts with the family and who initiated the contact; the duration of all contacts; the location of the contact; and the topic discussed, support provided, or toolkits reviewed.
Retention Rate | 9 months
  The number of families retained will be determined by the number of families who complete treatment Phase 2
Number of subjects consented | 9 months
  The number of families consented will be measured by the percentage of eligible families consenting to the study
Changes (or Improvement) with interpersonal relationships | 9 months
  This is a nine-item measure designed to assess satisfaction with the interpersonal relationship with the navigator or SW. The measure has been shown to have high internal consistency and to be significantly correlated with overall satisfaction with care and not to be correlated with health literacy or patients' primary language
Changes in ABC-irritability subscale | 6 months
  To meet eligibility the caregiver completed Aberrant Behavior Checklist-2 (ABC-2) Irritability subscale score needs to be > 13 (above the 50th percentile for children with ASD).This change will be measured by comparing the first stage interventions (SW vs. ABHN) and the change in ABC-irritability subscale score between baseline and the intermediate visit at month 3. At month 3, patients whose ABC Irritability subscale scores demonstrate improvement of at least 5 points (approximately ½ SD; moderate effect size) will remain in the same intervention. Patients whose ABC Irritability subscale scores suggest minimal to no improvement (less than 5 point improvement) will be randomized to either ABHN or ABHN+CAP if they were in the social work group in Phase 1 or will receive ABHN+CAP if they were in the ABHN arm of the study in phase 1. The primary efficacy endpoint for comparing the three embedded regimes will be ABC-irritability subscale at month 6.
Changes in levels of challenging behavior | 6 months
  This will be measured by the Clinician Global Impression Scales (CGI). The CGI consists of a severity scale (CGI-S) and an Improvement scale (CGI-I). For the CGI-I, clinicians use record review to rate the level of change from the screening/baseline visit (1-3 indicating improvement, 4 indicating no change, 5-7 indicating a worsening of symptoms). The CGI-I will be completed at the 3- and 6-month follow up visits, and will measure the level of improvement compared to the CGI-S taken at screening/baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan J Blum, M.D, Principal Investigator — Children's Hospital of Philadelphia; Judith S Miller, Ph.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Adams JS, Woods ER. Redesign of chronic illness care in children and adolescents: evidence for the chronic care model. Curr Opin Pediatr. 2016 Aug;28(4):428-33. doi: 10.1097/MOP.0000000000000368. PMID 27138998
- [Background] Bearss K, Johnson C, Smith T, Lecavalier L, Swiezy N, Aman M, McAdam DB, Butter E, Stillitano C, Minshawi N, Sukhodolsky DG, Mruzek DW, Turner K, Neal T, Hallett V, Mulick JA, Green B, Handen B, Deng Y, Dziura J, Scahill L. Effect of parent training vs parent education on behavioral problems in children with autism spectrum disorder: a randomized clinical trial. JAMA. 2015 Apr 21;313(15):1524-33. doi: 10.1001/jama.2015.3150. PMID 25898050
- [Background] Chakraborty B, Murphy SA. Dynamic Treatment Regimes. Annu Rev Stat Appl. 2014;1:447-464. doi: 10.1146/annurev-statistics-022513-115553. PMID 25401119
- [Background] Guinchat V, Cravero C, Diaz L, Perisse D, Xavier J, Amiet C, Gourfinkel-An I, Bodeau N, Wachtel L, Cohen D, Consoli A. Acute behavioral crises in psychiatric inpatients with autism spectrum disorder (ASD): recognition of concomitant medical or non-ASD psychiatric conditions predicts enhanced improvement. Res Dev Disabil. 2015 Mar;38:242-55. doi: 10.1016/j.ridd.2014.12.020. Epub 2015 Jan 7. PMID 25575287
- [Background] Johnson CR, DeMand A, Lecavalier L, Smith T, Aman M, Foldes E, Scahill L. Psychometric properties of the children's sleep habits questionnaire in children with autism spectrum disorder. Sleep Med. 2016 Apr;20:5-11. doi: 10.1016/j.sleep.2015.12.005. Epub 2015 Dec 29. PMID 27318219
- [Background] Linn KA, Laber EB, Stefanski LA. iqLearn: Interactive Q-Learning in R. J Stat Softw. 2015 Feb;64(1):i01. doi: 10.18637/jss.v064.i01. Epub 2015 Mar 20. PMID 26900385
- [Background] Shea S, Turgay A, Carroll A, Schulz M, Orlik H, Smith I, Dunbar F. Risperidone in the treatment of disruptive behavioral symptoms in children with autistic and other pervasive developmental disorders. Pediatrics. 2004 Nov;114(5):e634-41. doi: 10.1542/peds.2003-0264-F. Epub 2004 Oct 18. PMID 15492353
- [Background] Laurent PA. The emergence of saliency and novelty responses from Reinforcement Learning principles. Neural Netw. 2008 Dec;21(10):1493-9. doi: 10.1016/j.neunet.2008.09.004. Epub 2008 Sep 25. PMID 18938058
- [Background] Volker MA, Lopata C, Smerbeck AM, Knoll VA, Thomeer ML, Toomey JA, Rodgers JD. BASC-2 PRS profiles for students with high-functioning autism spectrum disorders. J Autism Dev Disord. 2010 Feb;40(2):188-99. doi: 10.1007/s10803-009-0849-6. Epub 2009 Aug 25. PMID 19705267